CLINICAL TRIAL: NCT04072497
Title: A Safety and Immunogenicity Study of a Zoster Vaccine in Healthy Adults >= 40 Years
Brief Title: A Clinical Study of a Zoster Vaccine in Healthy Adults >= 40 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017L04524-Ⅰ/Ⅱ
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Herpes Zoster
Keywords: VZV
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zoster vaccine, Live (Experimental): live attenuated varicella-zoster virus vaccine (with live virus >=4.3 LgPFU per dose)
  Interventions: Biological: One shot of the zoster vaccine
- Varicella vaccine, Live (Active Comparator): live attenuated varicella-zoster virus vaccine (with live virus >=3.3 LgPFU per dose)
  Interventions: Biological: One shot of the varicella vaccine
- Placebo (Placebo Comparator): Placebo with no live virus
  Interventions: Biological: one shot of placebo

INTERVENTIONS:
Biological: One shot of the zoster vaccine — One shot of the zoster vaccine (with live virus >=4.3 LgPFU per dose)
  Arms: Zoster vaccine, Live
Biological: One shot of the varicella vaccine — One shot of the varicella vaccine (with live virus >=3.3 LgPFU per dose)
  Arms: Varicella vaccine, Live
Biological: one shot of placebo — one shot of placebo with no live virus
  Arms: Placebo

SUMMARY:
Varicella-zoster virus (VZV) is a herpesvirus that causes two distinct clinical syndromes.Primary infection is manifested as varicella (chickenpox), whereas reactivation of latent VZV results in a localized eruption known as herpes zoster. Most people 40 years of age or older had evidence of previous VZV infection. This study plans to have 522 adults above 40 years old involoved in a randomized, double-blind, placebo-controlled trial of an investigational live attenuated zoster vaccine. The investigational vaccine is produced by Shanghai Institute of Biological Products Co., Ltd. The safety and immunogenicity of the zoster vaccine is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged over 40 years (male or female).
* Able to comply with all clinical trial protocol requirements and willing to complete all the visit plan process during the whole clinical trial observation period.
* Able to understand the content of informed consent and willing to sign the informed consent.
* Able to complete the diary card independently.
* Patients with chronic diseases need to be in a stable period.
* Axillary temperature ≤37.0°C.

Exclusion Criteria:

* Prior history of herpes zoster.
* Prior history of vaccination with herpes zoster vaccine or chickenpox vaccine.
* History of allergic disease likely to be exacerbated by any component of the vaccine.
* Taking immunoglobulins and/or any blood products within the last 3 months or will receive these products during the study period.
* Taking certain pharmaceuticals to be like salicylate kind, including aspirin, and difluorosalicylic, or going to take these medicine during the study period.
* Participation in another research study involving receipt of an investigational product in the last 30 days.
* Prior administration of live vaccine in last 30 days.
* Prior administration of subunit vaccine, inactivated vaccine or allergic therapy in last 14 days.
* History of serious disease and the participation in the clinical trial is likely to increase the disease risk and interfere with the observation of clinical trial index.
* Taking immunosuppressive therapy in last 6 months.
* Any autoimmune disease or immunodeficient state, autoimmune disease or immunodeficient disease.
* Active tuberculosis patient.
* Acute or chronic infections at the vaccination day (axillary temperature≥ 38.0°C).
* Coagulation disorders (coagulation factor deficiency, coagulopathy or platelet disorder) diagnosed by doctors, or obvious bruises or blood coagulation noticed.
* Woman who is breast-feeding.
* Previous history of mental and neurological diseases (e.g. depression, epilepsy or convulsion)
* Planned to move before the end of the study or leave the country for a long time during the scheduled study visit.
* Abnormal Blood Routine and Biochemical Indexes before Inoculation (except for minor abnormalities that are not clinically significant as judged by doctors)
* Any other conditions may compromise the safety or availability of participants in the judgment of the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Reactogenicity in the group of live attenuated zoster vaccine | 0 days-6 months after the vaccination
  * The incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * The incidence rate of subjects with solicited SAE(s) with 95% confidence interval
VZV specific serum conversion rate | 30 days after the vaccination
  VZV specific serum conversion is defined as: if serum antibody titer before immunization was less than 1: 8, and antibody titer after immunization was ≥ 1: 8. Or the antibody titer before immunization was≥1:8, and the antibody titer after immunization≥4-fold increase.
VZV specific serum geometric mean titre | 30 days after the vaccination
  For each group serum titre with FAMA test
VZV specific serum geometric mean fold increase | 30 days after the vaccination
  For each group serum titre with FAMA test

SECONDARY OUTCOMES:
Reactogenicity in the group of live attenuated varicella vaccine | 0 days-6 months after the vaccination
  * The incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * The incidence rate of subjects with solicited SAE(s) with 95% confidence interval
Reactogenicity in the group of placebo | 0 days-6 months after the vaccination
  * The incidence rate of subjects with solicited AE(s) with 95% confidence interval
  * The incidence rate of subjects with solicited SAE(s) with 95% confidence interval
The immunogenicity persistence of antibody titer | 90 days-360 days after vaccination
  The antibody titer measured by FAMA postvaccination in day 90,180,360

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial Center for Disease Control and Prevention, Zhaoge, Henan, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT04072497/Prot_SAP_000.pdf